CLINICAL TRIAL: NCT05491720
Title: Comparable Efficacy of Transcranial Direct Current Stimulation and Pharmacological Treatments in Children With Autism Spectrum Disorder
Brief Title: Electrical Brain Stimulation and Pharmacological Treatments in Autism Spectrum Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Brain Mapping Laboratory (NBML) (Other)
Collaborators: Ardabil University of Medical Sciences (Other); Leibniz Research Centre for Working Environment and Human Factors (Other); University of Tehran (Other)
Responsible Party: Principal Investigator, Mohammad Ali Salehinejad, Principal Investigator, The National Brain Mapping Laboratory (NBML)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.ARUMS.REC.1395.20
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Risperidone; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tDCS group (Experimental): TDCS intervention protocol consists of 10 sessions of 20 minutes of 1.5 mA electrical stimulation on consecutive days. Anodal electrode will be placed over the left dorsolateral prefrontal cortex and cathodal electrode will be placed over the right supraorbital area.
  Interventions: Device: transcranial direct current stimulation; Drug: Placebo
- Medication group (Experimental): Participants in this group will receive two daily Risperidone 1 mg tablets (Sobhan Pharmaceutical Company) for 10 consecutive days
  Interventions: Drug: RisperiDONE 1 MG/ML; Device: sham transcranial direct current stimulation
- Control group (Placebo Comparator): Participants in this group undergo 10 daily sessions of sham tDCS concurrent with placebo tablets ( Galenus pharmaceutical company) for 10 consecutive days.
  Interventions: Drug: Placebo; Device: sham transcranial direct current stimulation

INTERVENTIONS:
Drug: RisperiDONE 1 MG/ML — Patients will receive two daily Risperidone 1 mg tablets (Sobhan Pharmaceutical Company) for 10 consecutive days
  Arms: Medication group
Device: transcranial direct current stimulation — Patients will receive 10 sessions of 20 minutes of 1.5 mA electrical stimulation on consecutive days
  Other Names: tDCS
  Arms: tDCS group
Drug: Placebo — Patients will receive placebo tablet (Galenus pharmaceutical company)
  Arms: Control group; tDCS group
Device: sham transcranial direct current stimulation — Patients will receive 10 sessions of 20 minutes of sham electrical stimulation on consecutive days
  Arms: Control group; Medication group

SUMMARY:
This project aims to comparing the effectiveness of transcranial direct current stimulation with common pharmacological treatments on behavioral problems and cognitive deficits of children with autism spectrum disorder

DETAILED DESCRIPTION:
45 children with autism spectrum disorder are recruited in Fatemi Hospital at Ardabil University of Medical Sciences. The patients will be randomized into 3 Intervention groups of 15 with tDCS stimulation, risperidone, and placebo medication as the interventions. The study will be a randomized double-blind controlled design. The experimenter and the patient are blinded and are not aware of the study. Intervention group 1: TDCS intervention protocol consists of 10 sessions of 20 minutes of 1.5 mA electrical stimulation on consecutive days. Anodal electrode will be placed over the F3 and cathodal electrode will be placed over the Fp2. They will also receive a placebo tablet (Galenus pharmaceutical company) in each stimulation session. Intervention group 2: Participants in this group will receive two daily Risperidone 1 mg tablets (Sobhan Pharmaceutical Company) for 10 consecutive days. Intervention group 3: Participants in this group undergo 10 daily sessions of sham tDCS concurrent with a placebo tablet (Galenus pharmaceutical company) for 10 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder by a psychiatrist and behavioral checklist
* being 6-16 years old
* providing written informed consent signed by parents

Exclusion Criteria:

* comorbidity with other neurodevelopmental disorders
* comorbidity with other neurological disorders
* previous history of neurosurgery
* presence of any ferromagnetic metal in the head
* implanted medical devices in the head or neck region
* history of noncontrolled epilepsy with seizures in the last year

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Gilliam Autism Rating Scale (GADS) | up to 3 months after the intervention
  Score in the Gilliam Autism Rating Scale (GADS)
  Autism index scores:
  69 or less = unlikely 70-84 = possible 85 or higher = very likely
verbal fluency task | up to 3 months after the intervention
  Performance in the verbal fluency task as an executive and language function task
Theory of mind | up to 3 months after the intervention
  Score in the Theory of Mind Test (ToMT) Score range of subscales 1 to 3, is 0-20, 0-13, and 0-5, respectively and the total score range is 0-38.

CONTACTS AND LOCATIONS:
Locations (1):
- The National Brain Mapping Laboratory (NBML), Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided